CLINICAL TRIAL: NCT04169594
Title: Guiding Best Practice Clinical Care With In-Silico Rehabilitation and Statistical Parametric Mapping (SPM 1D) for Unilateral Chronic Hemiparetic Stroke and Trans-tibial Amputation: An Exploratory Clinical Study
Brief Title: Statistical Parametric Mapping (SPM 1D) for Stroke and Trans-tibial Amputation
Status: Completed | Type: Observational
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Nanyang Technological University (Other)
Responsible Party: Sponsor
Other Study IDs: DSRB_2019_99879
Record Dates: First submitted 2019-11-10; First posted 2019-11-20 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Stroke; Amputation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke: Unilateral hemiplegic stroke patients
  Interventions: Diagnostic Test: 3D Gait Analysis with Statistical Parametric Mapping
- Amputee: Unilateral transtibial amputee patients
  Interventions: Diagnostic Test: 3D Gait Analysis with Statistical Parametric Mapping

INTERVENTIONS:
Diagnostic Test: 3D Gait Analysis with Statistical Parametric Mapping — A 3D motion capture system will be used for gait analysis. Vector field statistics will be used to simplify the clinical interpretation of time varying movement patterns.

SUMMARY:
Gait analysis is commonly performed in clinical practice. However, it is complex and requires an understanding of the activation of muscles in lower limbs, trunk, and upper limbs in a specific spatiotemporal pattern and the appropriate joint positions which support and advance the body weight in different phases of gait cycles.

In study, we plan to pilot the application of 3D gait analysis with statistical modelling in 2 common causes of gait deviation: unilateral hemiplegic stroke and unilateral lower limb amputation.

DETAILED DESCRIPTION:
This is a pilot study on the use of 3D gait analysis using motion capture in combination with Statistical Parametric Mapping in patients with unilateral hemiplegic stroke and unilateral lower limb amputation. Data collected will then be compared against a normative dataset.

The findings from this study will then be used to build a decision support tool in combination with clinical analysis which could focus clinical recommendations for gait training, physical therapy, exercise and orthotics prescription to reduce unnecessary joint forces in affected and unaffected segments.

ELIGIBILITY:
Inclusion Criteria for stroke patients:

* First ever chronic unilateral hemiparetic stroke subjects, with stroke diagnosed by a physician and confirmed via CT/MRI
* >6 months post stroke
* ambulant with at most contact guard/standby supervision with/without walking aid during the study
* 10m Walk Test >/=0.2m/s and 6min Walking test walking distance of >/=50m without rest stop, with Functional Ambulation Category of >/=4 ((Holden et al, 1994)
* AMT>6
* able to understand study procedures and sign informed consent
* able to attend a single 2.5h session of research data collection.

Inclusion Criteria for amputee patients:

* First ever chronic unilateral transtibial amputee subjects
* intact residual limb
* > 6 months post amputation
* ambulant with at most contact guard/standby supervision with/without walking aid during the study
* 10m Walk Test >/=0.2m/s and 6min Walking test walking distance of >/=50m without rest stop
* with Medicare K level of >1
* AMT>6
* able to understand study procedures and sign informed consent
* able to attend a single 2.5h session of research data collection.

Exclusion Criteria:

* Unstable recent cardiorespiratory conditions including uncontrolled hypertension/ hypotension, angina pectoris, myocardial infarction, active congestive cardiac failure, untreated cardiac arrhythmias (e.g. atrial fibrillation), untreated pulmonary embolism or deep vein thrombosis, presence of cardiac pacemaker.
* Functional status: severe aphasia or neglect (inability to obey 1 steps command), communication disorder precluding understanding of instructions, cognitive impairment, dementia, untreated depression or psychiatric disorder.
* End stage conditions such as medical instability or orthostatic insufficiency, organ, renal, liver, heart failure and life expectancy <6 months or on haemodialysis.
* Pregnancy.
* Local limb conditions which could be exacerbated by research interventions such as open wounds, ulcers, stump pain or stump wounds/ulcers, neuromas in amputees, active arthritis or joint or limb pain.
* Skin conditions which could be worsened by application of adhesive skin markers such as uncontrolled eczema, psoriasis, fungal or bacterial infections etc.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients in outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Body movement assessed by a motion capture system | Assessed within 1 year after patient recruitment
  Direction and magnitude of each body movement will be combined to provide graphical data on a motion capture system

SECONDARY OUTCOMES:
Fugl Meyer Assessment | Assessed within 1 year after patient recruitment
  Functional score for stroke patients. Minimum: 0, Maximum: 226, with higher score indicating better function
Stroke Impact Scale | Assessed within 1 year after patient recruitment
  Functional score for stroke patients. Minimum:1, Maximum: 5, with higher score indicating higher impairment
Amputee Mobility Predictor with prosthesis | Assessed within 1 year after patient recruitment
  Functional score for amputation patients. Minimum: 0, Maximum: 47, with higher score indicating better function.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Chua, Principal Investigator — Tan Tock Seng Hospital; Cyril Donnelly, Principal Investigator — Rehabilitation Research Institute of Singapore
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No